CLINICAL TRIAL: NCT02215070
Title: Prevention of Gastrointestinal Toxicity From Total Body Irradiation or High Dose Chemotherapy With Pasireotide
Brief Title: Pasireotide in Prevention of GI Toxicity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anthony Sung, MD (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, Anthony Sung, MD, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00051736
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Results first posted 2020-03-11 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: Hematological Malignancies
Keywords: Allogeneic Stem Cell Transplantation; Acute Myeloid Leukemia; Acute Lymphoid Leukemia; Acute Non-Lymphocytic Leukemia; Myelodysplastic Syndrome; Chronic Myeloid Leukemia; Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pasireotide + Preparatory Regimen (Experimental): Eligible subjects will receive pasireotide daily for 5 days before stem cell transplant, the day of the stem cell transplant, and daily for 8 days following the stem cell transplant. Preparatory regimen will be given 4 days before stem cell transplant.
  Interventions: Drug: Pasireotide

INTERVENTIONS:
Drug: Pasireotide — Eligible subjects will receive pasireotide daily for 5 days before stem cell transplant, the day of the stem cell transplant, and daily for 8 days following the stem cell transplant. Preparatory regimen will be given 4 days before stem cell transplant.

SUMMARY:
The purpose of this study is to evaluate if the drug, Pasireotide, is safe and effective in reducing the gastrointestinal side effects of the drugs received to prepare for allogeneic stem cell transplant. The study will also evaluate if Pasireotide is effective in reducing acute and chronic Graft-versus-Host-Disease (GvHD) after transplant.

DETAILED DESCRIPTION:
The study design will be a non-randomized phase II. Forty patients receiving an ablative preparatory regimen will receive pasireotide subcutaneous (0.9 mg, b.i.d.) one day prior to initiation of the preparatory regimen and continuing for eight days following the completion of the preparatory regimen not to exceed 14 days total dosing. We select matched controls from existing patients who did not take the drug to minimize the time it takes to complete the trial.

Myeloablative preparatory regimens are defined as those including either TBI ≥ 1200 cGy or busulfan ≥ 12.8 mg/kg. The most common regimens combine TBI with cyclophosphamide (TBI/Cy) or busulfan with cyclophosphamide (Bu/Cy) (Appendix E). However, any regimen meeting the above definition of myeloablative preparatory regimen may be used.

The study will collect data at screening, at baseline prior to initiation of the drug (day of study drug start), transplant day 0, day +7, day +14 and weekly thereafter until day +100, and on days +180, +270, and +365. The total days on pasireotide therapy will be recorded as well as any SAE that is outside the expected for stem cell transplantation. We will also follow the incidence and severity of acute and chronic GVHD.

At Duke only, a video capsule endoscopy will be performed in a subset of ten study patients between transplant days +4 through +6. This substudy is descriptive in nature and only used to collect a source of preliminary data that may suggest further study.

Patients must agree to participate in this portion of the study and will be asked to sign a clinical consent for performance use of the video capsule endoscopy. Patients will be given detailed instructions to prepare for the procedure. An investigator who is blinded to the group allocation of the patients/volunteers separately will review the images obtained from each of the capsule examinations. Images will be examined for evidence of the four following types of abnormalities: reddened/edema/villous blunting, erosion, ulcer and stenosis. Each of these categories will be scored from 0-3 and summed to obtain an overall index that will range from 0 (normal study) to 12 (severely abnormal in all categories).

Citrulline assay Measurement of citrulline concentration has been used as a marker for cytotoxic treatment-induced intestinal damage and it is highly reproducible. The citrulline concentration appears to be a quantitative parameter that is independent of the underlying cause for epithelial cell loss and functions well in the post-SCT setting. Six mls of blood will be collected in heparinized tubes on days 0, 7, and 14. Tubes will be centrifuged according to manufacturer's instructions and the plasma will be collected and stored at -80C until shipment to the laboratory performing the assay.

Calprotectin assay Calprotectin has been described as another biomarker of GI injury. During radiation-induced inflammation, leucocytes infiltrate the mucosa and increase the level of fecal calprotectin. At least 50 mg of stool specimen will be collected from patients on days 0, 7, and 14. Samples will be stored at -80C until shipment to the laboratory performing the assay. Calprotectin will be measured with an ELISA kit (CALPRO, Oslo, Norway) in accordance with the manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at the time of study enrollment.
* Histologically confirmed diagnosis for which an allogeneic transplant is utilized.
* Plan to receive an allogeneic transplant from a 4-6/6 single or dual umbilical cord blood graft, or a 7-8/8 HLA-matched sibling or unrelated donor (High resolution HLA-A, B, C, DRB1).
* Meet standard criteria as defined by the institution for a myeloablative allogeneic stem cell transplantation, with myeloablative defined as using conditioning regimens containing:

  * TBI ≥ 1200 cGy, or
  * Busulfan ≥ 12.8mg/kg
* Patient must have given written informed consent according to FDA guidelines.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.

Exclusion Criteria:

* Female patients who are pregnant or lactating, or are of childbearing potential (FCBP, defined as all women physiologically capable of becoming pregnant) and not practicing an effective method of contraception/birth control
* FCBP must have a current negative serum pregnancy test prior to transplant per institutional practice.
* Use of an investigational drug within 1 month prior to dosing. Concurrent enrollment on other clinical research studies that contain an interventional therapy is not permitted while subjects are receiving pasireotide or within 5 half-lives of finishing pasireotide. However, subjects may concurrently enroll in non-interventional studies (e.g. biobanking, mobile health tracking).
* Active CNS disease (related to primary malignancy) at the time of enrollment.
* Patients with existing grade 2 toxicities, except as approved by the investigator.
* Any of the following diseases or conditions:

Cardiac:

* History of unexplained syncope or family history of idiopathic sudden death.
* Sustained or clinically significant cardiac arrhythmias.
* Risk factors for Torsades de Pointes such as:

  * Uncontrolled hypokalemia
  * Uncontrolled hypomagnesemia or hypermagnesemia
  * Cardiac failure (New York Heart Association Class II or higher)
  * Clinically significant/symptomatic bradycardia (HR < 50), or high-grade AV block.
  * Known diagnosis of QT prolongation (QTc ≥ 470) or family history of long QT syndrome
  * Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes, or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism or cardiac failure.
  * Concomitant medications known to prolong the QT interval during the same time as pasireotide is to be administered (unless approved by PI and QTc < 470; standard transplant medications that are known to prolong the QT (e.g. azoles, ondansetron, etc.) are permitted but caution is advised and patients should be closely monitored).

Endocrine:

* Uncontrolled diabetes at the time of cytoreduction. All patients with diabetes must be optimized on their diabetes regimen prior to initiating pasireotide.

  • If a patient is diabetic: uncontrolled diabetes as defined by HbA1c > 8 per cent despite adequate therapy
* Patients who are not biochemically euthyroid. Patients with known history of hypothyroidism are eligible if they are on adequate and stable replacement thyroid hormone therapy for at least 3 months.
* Known diagnosis of hypocortisolism
* Known diagnosis of pituitary hormone deficiency.
* Known hypersensitivity to somatostatin analogs or any component of the pasireotide LAR or s.c. formulations.

Infectious:

* Uncontrolled (not being treated) infections at the time of cytoreduction.
* A positive HIV test result (ELISA and Western blot) or history of known HIV. An HIV test will not be required; however, previous medical history will be reviewed.

Gastrointestinal:

* Moderately impaired hepatic function (Child-Pugh B) or severe hepatic impairment (Child-Pugh C)
* Known gallbladder or bile duct disease, symptomatic cholelithiasis, acute or chronic pancreatitis.
* Known malabsorption syndrome, short bowel or chologenic diarrhea not controlled by specific therapeutic means.

Hematologic:

* Abnormal coagulation (PT or aPTT > 30% above normal limits).
* Continuous anticoagulation therapy. Patients who were on anticoagulant therapy must complete a washout period of at least 10 days and have confirmed normal coagulation parameters before study inclusion.

Miscellaneous:

* Major surgery/surgical therapy for any cause within 1 month prior to pasireotide administration. Patients should have recovered and have a good clinical condition before entering the study.
* Any co-morbid condition which, in the view of the Principal Investigator, renders the patient at high risk from treatment complications.

Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Sung, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 enrolled participants screen failed, 5 withdrew, and 1 was withdrawn by physician decision.
Groups:
- Historical Controls: Contemporaneous controls were matched using the following parameters: Transplant diagnosis (acute leukemias, lymphomas, myelodysplastic syndrome [MDS]/myeloproliferative neoplasm [MPN]/other), donor (related, unrelated), graft (bone marrow, peripheral blood progenitor cell [PBPC], and cord), GVHD prophylaxis (tacrolimus/methotrexate), age, hematopoietic cell transplantation-specific comorbidity index (HCT-CI), and conditioning regimen (TBI-based, chemotherapy only).
Period: Overall Study
Arm/Group | Pasireotide + Preparatory Regimen | Historical Controls
Started | 26 | 52
Completed | 20 | 52
Not Completed | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pasireotide + Preparatory Regimen | Historical Controls | Total
Number analyzed (Participants) | 26 | 52 | 78
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [41 to 62] | 51 [36 to 52] | 52 [40 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Gender: Female | 8 | 23 | 31
  Gender: Male | 18 | 29 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 26 | 46 | 72
  Unknown or Not Reported | 0 | 5 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 7 | 9
  White | 23 | 43 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 52 | 78

OUTCOME MEASURES:

1. Primary Outcome: Percentage of GI Toxicity From the Preparatory Regimen and the GVHD Prophylaxis in Stem Cell Transplantation (SCT) Patients Who Are Treated With Pasireotide
Description: Number of participants who experience grades III-IV GI toxicity
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Pasireotide + Preparatory Regimen
Number analyzed (Participants) | 26
Participants | 21

2. Secondary Outcome: Percentage of Acute GVHD
Description: Number of participants who experience acute GVHD
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pasireotide + Preparatory Regimen
Number analyzed (Participants) | 26
Participants | 15

3. Secondary Outcome: Maximum Severity of Acute GVHD Compared to Historical Controls
Description: Assess maximum severity of acute GVHD scored as stage 1 (least severe) through stage 4 (most severe) using BMT CTN, 2013 standards
Time Frame: 100 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Pasireotide + Preparatory Regimen
Number analyzed (Participants) | 26
units on a scale | 2 [1 to 3]

4. Secondary Outcome: Incidence of Chronic GVHD Compared to Historical Controls
Description: Measure the number of participants who experience chronic GVHD
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pasireotide + Preparatory Regimen | Historical Controls
Number analyzed (Participants) | 26 | 52
Participants | 16 | 22
Statistical Analysis 1: Comparison: Pasireotide + Preparatory Regimen vs Historical Controls; Test type: Other; p = 0.12, Chi-squared

5. Secondary Outcome: Maximum Severity of Chronic GVHD Compared to Historical Controls
Description: Assess maximum severity of chronic GVHD scored as none, mild, moderate or severe using 2014 NIH Consensus Criteria
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pasireotide + Preparatory Regimen | Historical Controls
Number analyzed (Participants) | 26 | 52
Participants | 8 | 11

6. Secondary Outcome: Overall Survival Compared to Historical Controls
Description: Rate of overall survival of participants at one year post transplant
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pasireotide + Preparatory Regimen | Historical Controls
Number analyzed (Participants) | 26 | 52
percentage of participants | 63 [47 to 86] | 82 [72 to 93]
Statistical Analysis 1: Comparison: Pasireotide + Preparatory Regimen vs Historical Controls; Test type: Other; p = 0.006, Log Rank

7. Secondary Outcome: Disease Free Survival Compared to Historical Controls
Description: Rate of disease free survival of participants at one year post transplant
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pasireotide + Preparatory Regimen | Historical Controls
Number analyzed (Participants) | 26 | 52
percentage of participants | 40 [25 to 65] | 78 [68 to 91]
Statistical Analysis 1: Comparison: Pasireotide + Preparatory Regimen vs Historical Controls; Test type: Other; p = 0.002, Log Rank

8. Other Pre Specified Outcome: Citrulline and Fecal Calprotectin Levels Will be Measured
Description: Exploratory outcome-These levels will be evaluated as biomarkers of GI tract health and function in SCT patients and the correlation between these biomarkers and GI toxicity.
Time Frame: 100 days
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Evaluate GI Toxicity Assessment by Video Capsule Endoscopy.
Description: Exploratory outcome-Video capsule endoscopy will be performed in a subset of ten study participants on the last day study drug is administered. Images will be examined for evidence of the four following types of abnormalities: reddened/edema/villous blunting, erosion, ulcer and stenosis.
Time Frame: 14 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AEs were reported from the day Pasireotide started to day 30 after transplant (Day +30).
Description: Adverse event collection is not applicable for historical controls. Adverse events after Day 30 were not expected to be related to the intervention. However, HCT is a fraught process, with significant morbidity, and 10-20% of patients die from transplant-related complications. To determine if the study intervention would improve survival, overall survival was collected at year 1 (efficacy) and adverse events between Day 30-Year 1 were not collected.
Arm/Group | Pasireotide + Preparatory Regimen | Historical Controls
All-Cause Mortality (participants affected / at risk) | 1/26 | 0/0
Serious Adverse Events (participants affected / at risk) | 8/26 | 0/0
Other Adverse Events (participants affected / at risk) | 26/26 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide + Preparatory Regimen (N=26) | Historical Controls (N=0)
Mobitz - Type II AV Block (Cardiac disorders) | 1 | NA
Enterocolitis (Gastrointestinal disorders) | 1 | NA
VOD (Hepatobiliary disorders) | 1 | NA
Somnolence (Nervous system disorders) | 1 | NA
Febrile Neutropenia (Infections and infestations) | 2 | NA
Infections and infestations - Other, specify; blood stream (Infections and infestations) | 1 | NA
Lung infection (Infections and infestations) | 1 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide + Preparatory Regimen (N=26) | Historical Controls (N=0)
Abdominal Pain (Gastrointestinal disorders) | 14 | NA
Anorexia (Gastrointestinal disorders) | 21 | NA
Bloating (Gastrointestinal disorders) | 5 | NA
Constipation (Gastrointestinal disorders) | 8 | NA
Diarrhea (Gastrointestinal disorders) | 24 | NA
Dysphagia (Gastrointestinal disorders) | 1 | NA
Dyspepsia (Gastrointestinal disorders) | 5 | NA
Dysgeusia (Gastrointestinal disorders) | 9 | NA
Allergic reaction (Immune system disorders) | 2 | NA
Afib (Cardiac disorders) | 0 | NA
Anxiety (Psychiatric disorders) | 7 | NA
Chills (General disorders) | 1 | NA
Sinus Bradycardia (Cardiac disorders) | 7 | NA
2nd deg AVB (Cardiac disorders) | 1 | NA
Chest pain (General disorders) | 2 | NA
Enterocolitis (Infections and infestations) | 5 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | NA
Inreased Creatinine (Renal and urinary disorders) | 5 | NA
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | NA
Acute Kidney Injury (Renal and urinary disorders) | 0 | NA
Dry Eyes (Eye disorders) | 2 | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | NA
Epistaxis (General disorders) | 2 | NA
Dysuria (Renal and urinary disorders) | 6 | NA
Bone Pain (General disorders) | 1 | NA
Bladder Spasm (Renal and urinary disorders) | 1 | NA
Dehydration (General disorders) | 1 | NA
URI (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Myocardial Infarction (Cardiac disorders) | 0 | NA
Encephalopathy (Nervous system disorders) | 6 | NA
Fatigue (General disorders) | 20 | NA
Febrile Neutropenia (Infections and infestations) | 17 | NA
Fever (Infections and infestations) | 4 | NA
Floaters (Eye disorders) | 0 | NA
Fracture (General disorders) | 1 | NA
Folliculitis (Skin and subcutaneous tissue disorders) | 0 | NA
Hiccups (General disorders) | 0 | NA
Hallucination (Nervous system disorders) | 3 | NA
Headache (Nervous system disorders) | 11 | NA
Intracranial Hemorrhage (Nervous system disorders) | 0 | NA
Hematoma (Blood and lymphatic system disorders) | 0 | NA
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Hematuria (Renal and urinary disorders) | 1 | NA
HSV Reactivation (Infections and infestations) | 3 | NA
Hyperkalemia (Metabolism and nutrition disorders) | 3 | NA
Hypernatremia (Metabolism and nutrition disorders) | 1 | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 | NA
Hyperglycemia (Endocrine disorders) | 12 | NA
Hyponatremia (Metabolism and nutrition disorders) | 1 | NA
Hypertension (Vascular disorders) | 14 | NA
Hypotension (Vascular disorders) | 5 | NA
Infusion Reaction (Immune system disorders) | 3 | NA
Insomnia (General disorders) | 4 | NA
Lung Infection (Infections and infestations) | 4 | NA
Myalgias (General disorders) | 0 | NA
Nasal Congestion (General disorders) | 8 | NA
Otitis Media (Infections and infestations) | 1 | NA
Pain in Extremity (General disorders) | 1 | NA
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | NA
Pruritis (General disorders) | 2 | NA
Joint Infection (Infections and infestations) | 0 | NA
Menorrhagia (General disorders) | 0 | NA
Pericardial effusion (Cardiac disorders) | 1 | NA
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Pulmonary Edema (Cardiac disorders) | 4 | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | NA
Prostatic Obstruction (Renal and urinary disorders) | 1 | NA
Acne Rash (Skin and subcutaneous tissue disorders) | 1 | NA
Rhinorrhea (General disorders) | 3 | NA
Rash (Skin and subcutaneous tissue disorders) | 19 | NA
Skin Infection (Infections and infestations) | 3 | NA
Catheter-Related Infection (Infections and infestations) | 6 | NA
Toe Trauma (General disorders) | 1 | NA
PRES (Nervous system disorders) | 0 | NA
Sinusitis (Infections and infestations) | 0 | NA
Sepsis (Infections and infestations) | 7 | NA
Thromboembolic event (Blood and lymphatic system disorders) | 1 | NA
Thrush (Infections and infestations) | 4 | NA
Urinary incontinence (Renal and urinary disorders) | 1 | NA
UTI (Infections and infestations) | 2 | NA
Urinary Retention (Renal and urinary disorders) | 3 | NA
Viremia (Infections and infestations) | 4 | NA
VOD (Hepatobiliary disorders) | 1 | NA
AST Elevation (Hepatobiliary disorders) | 2 | NA
ALT Elevation (Hepatobiliary disorders) | 2 | NA
Alk Phos Elevation (Hepatobiliary disorders) | 1 | NA
Bilirubin Elevation (Hepatobiliary disorders) | 6 | NA
Mucositis (Gastrointestinal disorders) | 24 | NA
Ileus (Gastrointestinal disorders) | 2 | NA
Nausea (Gastrointestinal disorders) | 25 | NA
Vomiting (Gastrointestinal disorders) | 20 | NA
Bowel Obstruction (Gastrointestinal disorders) | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT02215070/Prot_SAP_000.pdf